CLINICAL TRIAL: NCT07047976
Title: A Study on the Mechanisms of Sulforaphane in Improving Autism Spectrum Disorder
Brief Title: Mechanism Study of Sulforaphane in ASD Improvement
Acronym: ASD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated prior to full implementation due to logistical and resource-related considerations. Study procedures and feasibility are currently being re-evaluated, and a revised protocol is under development for future implementation.
Sponsor: Jian-Jun Ou (Other)
Responsible Party: Sponsor-Investigator, Jian-Jun Ou, Principal investigator, Central South University
Organization: Central South University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYG20240055
Record Dates: First submitted 2025-02-10; First posted 2025-07-02 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Sulforaphane
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sulforaphane Intervention Group for Autism Spectrum Disorder (Experimental)
  Interventions: Dietary Supplement: Sulforaphane

INTERVENTIONS:
Dietary Supplement: Sulforaphane — This intervention involves the administration of Sulforaphane, a compound derived from glucoraphanin found in cruciferous vegetables. Participants will receive Avmacol® tablets, each containing 30 mg of glucoraphanin (approximately 68 μmol per tablet). They will take 3 tablets daily, resulting in a total daily dosage of approximately 90 μmol of Sulforaphane. The intervention will last for 8 weeks, during which participants will be monitored for clinical and biological outcomes.

SUMMARY:
The goal of this clinical trial is to find out if sulforaphane (SFN) can improve social skills and behavior in people with Autism Spectrum Disorder (ASD). ASD is a developmental disorder that affects how children and teenagers interact with others. The number of people diagnosed with ASD has been rising, putting a lot of pressure on families and society. The investigators hope this study will lead to new treatments.

The main questions the investigators want to answer are:

Can sulforaphane help improve social communication in people with ASD? How does sulforaphane affect the balance of certain chemicals in the brain?

The investigators will recruit 50 participants aged 12 to 34 diagnosed with ASD and 30 healthy volunteers for comparison. Participants will:

Take 3 capsules of sulforaphane each day for 8 weeks. Complete regular psychological tests, undergo brain scans, and have their brain activity monitored to assess the treatment's effectiveness.

Through this study, the investigators aim to discover the potential benefits of sulforaphane for individuals with ASD and provide new insights for future treatment options.

DETAILED DESCRIPTION:
This study aims to investigate the mechanisms by which sulforaphane (SFN) ameliorates the excitatory/inhibitory imbalance in patients with Autism Spectrum Disorder (ASD). ASD is a pervasive developmental disorder characterized by impairments in social communication, interaction, and stereotyped behaviors. In recent years, the prevalence of ASD has been rising, imposing a significant burden on families and society. Although current primary interventions focus on educational training, there is a lack of effective biological treatments. Preliminary studies have demonstrated that sulforaphane can safely and effectively improve core clinical symptoms in Chinese patients with ASD, showing significant associations with metabolites related to excitatory/inhibitory balance, such as taurine and phosphatidylserine.

This open-label study will recruit 50 ASD patients aged 12-34 years and 30 healthy controls for an 8-week clinical trial. The study will employ psychological and behavioral assessments, electroencephalography (EEG), and magnetic resonance imaging (MRI) to comprehensively evaluate changes in clinical phenotype and neurotransmitter levels in ASD patients. The primary outcome measure will be improvements in social communication, while secondary measures will include changes in other clinical symptoms and neurophysiological characteristics.

Through this study, the investigators aim to gain a deeper understanding of the effects of sulforaphane on ASD patients, providing a new theoretical foundation and clinical evidence for the precise treatment of ASD.

ELIGIBILITY:
Inclusion Criteria for ASD Group:

1. Age between 12-34 years.
2. Diagnosis of Autism Spectrum Disorder (ASD) as per the DSM-V criteria.
3. Diagnosis of ASD according to the Autism Diagnostic Interview-Revised (ADI-R).
4. Diagnosis of ASD based on the Autism Diagnostic Observation Schedule (ADOS).

Exclusion Criteria for ASD Group:

a. Presence of severe physical illnesses or conditions, such as:

1. Congenital heart disease
2. Thyroid disorders
3. Liver or kidney dysfunction
4. Visual or hearing impairments b. Severe neurological diseases with a clear family history or potential risk factors, such as:

a)Traumatic brain injury b) Encephalitis c) Epilepsy d) High fever seizures e) Birth trauma f） Abnormal EEG c. Known or suspected genetic disorders, such as:

1. Down syndrome
2. Fragile X syndrome d. Diagnosis of other developmental disorders, such as:

a) Isolated intellectual disability b) Isolated language development disorder c) Selective mutism e. Diagnosis of other major psychiatric disorders, such as:

1. Schizophrenia
2. Bipolar disorder f. Currently taking other psychiatric or neurological medications.

Inclusion Criteria for Healthy Control Group:

1. Age between 12-34 years.
2. No diagnosis of any mental disorders.

Exclusion Criteria for Healthy Control Group:Exclusion criteria are the same as those for the ASD group.

Ages: 12 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Social communication changes index | At baseline, week 4, and week 8
  Assessed by the Social Response Scale (SRS-II). This scale is used to evaluate the severity of social symptoms associated with autism spectrum disorders and includes five subdimensions: social awareness, social cognition, social communication, social motivation, and autism behaviors. The change in social communication scores from baseline to the end of the study period will be the primary outcome of interest. The critical value is 59.5, and the total score is the sum of all entries, with the lowest score of 0 and the highest score of 3 for each entry. The total score of this scale represents the severity of social functioning impairments in the participants, with higher scores indicating greater severity.
Autism assessment index | At baseline, week 4, and week 8
  Autism was assessed using the Oregon State University Autism Rating Scale, DSM-5 (OARS-5), which includes the signs and symptoms of autism spectrum disorders described in the DSM-5. The scores include :1; Total number of symptoms. Every symptom that occurs (i.e., 1, 2, or 3 points) is recorded in the symptom count. 2. Weighted average severity. The clinician scored each item on a scale of 0, 1, 2 or 3 based on the parent's description of the particular problem. 3. Damage index. In Section C of OARS-5, after discussion with the child/adolescent's caregiver, the clinician will rate the level of support on a scale of 0(no support) to 3(maximum support). In the OARS-5 scale, higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Functional E/I Ratio in EEG | At baseline, week 4, and week 8
  Detect resting state and task state EEG, analyze and calculate the functional E/I ratio.
Concentration Ratios of Neurotransmitters in Magnetic Resonance Spectroscopy | At baseline, week 4, and week 8
  The content and ratio of Glu/Cr, γ-GABA/Cr, NAA/Cr, Cho/Cr, and MI/Cr were detected by magnetic resonance spectroscopy to evaluate the changes in the key transmitters of neural E/I balance.
Eye Movement Parameters During Cognitive Tasks | At baseline, week 4, and week 8
  This outcome measure will utilize an eye tracker to record and analyze the visual movement trajectories of participants while they engage in cognitive tasks. The analysis will focus on the following parameters: (1) the fixation points, indicating what the participants look at during the tasks; (2) the frequency of fixations, reflecting how many times each visual target is observed; and (3) the duration of each fixation, representing how long participants focus on specific elements.
Performance on the 'Reading the Mind in the Eyes' Test | At baseline, week 4, and week 8
  The "Reading the Mind in the Eyes" test is a psychological assessment designed to measure a subject's ability to understand or infer the mental states of others through the observation of their eyes. It is used to investigate social cognition, empathy, and theory of mind. The test consists of 36 images, and for each image, participants receive one point if they correctly identify the mental state being expressed; otherwise, they receive zero points. A higher score indicates a greater proficiency in understanding others' mental states through facial cues.
Score on the Frith-Happe Animations Task | At baseline, week 4, and week 8
  The Frith-Happe animations task is used to measure individuals' ability to understand and interpret social interactions. In this task, participants are shown 8 short animated video clips depicting simple social interactions between triangle shapes. Participants will be asked whether the type of interaction of triangles in these animations is random or psychological, and be rated according to their choice of the type of interaction presented by the triangle animation. Each animation gets one point if it chooses the interaction type correctly; otherwise, it gets zero points. The total score is eight.
Score on the Strange Stories Task | At baseline, week 4, and week 8
  Strange Stories Task involves presenting participants with a series of short narrative vignettes that involve interactions between characters that require the reader to infer the characters' thoughts, beliefs, intentions, and emotions. After reading each story, participants are asked questions or prompted to make judgments about the characters' mental states, motivations, and interpretations. Responses are then scored based on the participant's ability to accurately interpret the social cues presented in the narratives. Each question is scored 0, 1, and 2 according to the scoring standard.
Clinical global impression assessment index | At baseline, week 4, and week 8
  The Clinical Global Impression Scale (CGI) is utilized to evaluate clinical efficacy. It consists of three components: Severity of Illness (SI), Global Improvement (GI), and Efficacy Index (EI). Each component uses an 8-point scale from 0 to 7, where 0 indicates no issues and 7 reflects the most severe condition. The total scores help clinicians assess the severity of the patient's condition, the degree of improvement or worsening from baseline, and the overall efficacy of the treatment considering both its effects and side effects. Higher scores generally indicate greater severity or deterioration, while lower scores suggest better outcomes.
Assessment of treatment outcomes in autism spectrum disorder | At baseline, week 4, and week 8
  The Autism Treatment Evaluation Checklist (ATEC) is used to assess changes in the severity of Autism Spectrum Disorder (ASD) in children aged 2 to 12 years following treatment. The ATEC consists of four sections: I. Expression/Language Communication (14 items), II. Social Skills (20 items), III. Perception/Cognitive Skills (18 items), and IV. Health/Behavior (25 items). The scores from each subscale are combined to calculate a total score, which ranges from 0 to 179. The initial assessment score is referred to as the 'baseline total score,' with mild (baseline ATEC total score 20-49), moderate (baseline ATEC total score 50-79), and severe (baseline ATEC total score >80) classifications. A lower score indicates milder severity of ASD. The primary purpose of the ATEC is to evaluate individual changes following interventions by comparing the baseline ATEC score with subsequent scores.
Adult ADHD symptom assessment index | At baseline, week 4, and week 8
  The Adult Self-Report Scale (ASRS) and the Wender Utah Rating Scale (WURS) are self-report tools for adults to assess Attention Deficit Hyperactivity Disorder (ADHD) symptoms.
  The ASRS has 18 questions covering two dimensions: attention deficits and hyperactive/impulsive behavior. Responses are rated on frequency using options like 'never,' 'rarely,' 'sometimes,' 'often,' or 'very frequently.' Each item scores from 0 (no problem) to 4 (most severe). The total ASRS score is the sum of all item scores.
  The WURS consists of 15 questions assessing childhood symptoms related to ADHD that may persist into adulthood. Responses are rated similarly, with options like 'not at all or very rarely,' 'rarely,' 'sometimes,' 'often,' or 'very often.' Each item scores from 0 to 4, with the total WURS score reflecting the severity of ADHD symptoms.
Adult executive functioning assessment index | At baseline, week 4, and week 8
  The Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) is a standardized measure designed to assess executive functioning and self-regulation in adults within everyday environments. It utilizes both self-report and informant-report formats. The scale comprises 75 items across 9 theoretically and empirically derived clinical scales: inhibition, self-monitoring, planning/organization, shifting, initiation, task monitoring, emotional control, working memory, and material organization. Responses are typically rated based on frequency, with options such as 'never,' 'occasionally,' and 'often.' Each item is scored on a scale from 1 to 3, where 1 indicates no problem and the highest score reflects the most severe problem. The total score of the BRIEF-A is the sum of the scores of all items, providing an overall assessment of executive function difficulties.
Depressive symptoms assessment index | At baseline, week 4, and week 8
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used clinical tool for assessing depressive symptoms. Based on the diagnostic criteria of the American Psychiatric Association, it helps clinicians screen for, diagnose, and evaluate the treatment effects of depression by asking patients about their depressive symptoms over the past two weeks. The scale consists of 9 items, with responses typically rated based on frequency and duration options such as 'not at all,' 'several days,' 'more than half the days,' and 'nearly every day.' Each item is scored on a scale from 0 to 3, where 0 indicates no problem and the highest score reflects the most severe symptoms. The total score of the PHQ-9 is the sum of all item scores, providing an overall assessment of depressive symptom severity.
Anxiety symptoms assessment index | At baseline, week 4, and week 8
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a self-assessment tool used to evaluate anxiety symptoms. The scale consists of 7 items that assess various aspects of anxiety. Responses are typically rated based on frequency and duration options such as 'not at all,' 'several days,' 'more than half the days,' and 'nearly every day.' Each item is scored on a scale from 0 to 3, with 0 indicating no problem and the highest score reflecting the most severe symptoms. The total score of the GAD-7 is the sum of all item scores, providing an overall assessment of anxiety symptom severity.
Manic symptoms assessment index | At baseline, week 4, and week 8
  The Altman Self-Rating Mania Scale (ASRM) is a diagnostic tool designed to assess the presence and severity of manic symptoms in individuals. The scale consists of 5 questions that evaluate various aspects of mania. Responses are typically rated based on frequency and duration options such as 'none,' 'occasionally,' 'often,' 'most of the time,' and 'nearly every day.' Each item is scored on a scale from 0 to 4, with 0 indicating no problem and the highest score reflecting the most severe symptoms. The total score of the ASRM is the sum of all item scores, providing an overall assessment of manic symptom severity.
Cross-Cutting symptom assessment index | At baseline, week 4, and week 8
  The Cross-Cutting Symptom Measures, developed by the DSM-5 Working Group, is a self-report tool for dimensional evaluation of adult patients' mental symptoms. It encompasses 13 dimensions and 23 items, including depression, anger, anxiety, and substance use. Ratings are based on frequency and duration, using a scale from 'not at all' to 'nearly every day.' Each item is scored from 0 (no problem) to 4 (most severe), with the total score reflecting the overall symptom severity.
Camouflaging behavior assessment index | At baseline, week 4, and week 8
  Camouflaging Autistic Traits Questionnaire (CAT-Q) is used to assess social camouflaging behaviors in adults. The questionnaire consists of 25 items, covering three dimensions: compensation, masking, and blending in, which reflect different social camouflage strategies. Ratings are based on a scale from 1 to 7, indicating the severity of behaviors. Higher scores indicate a greater level of social camouflaging, suggesting that individuals may engage in more camouflage behaviors in their daily lives; lower scores suggest less camouflage behavior, which may be associated with a more natural social approach.
Borderline symptom severity index | At baseline, week 4, and week 8
  The Borderline Symptom List 23 (BSL-23) is a self-assessment scale used to measure the extent of intrapsychic stress in patients with borderline personality disorder. The BSL-23 consists of three parts: 23 items that assess the individual's mental state over the past week, a visual analog scale to evaluate current mental well-being, and a supplementary scale with 11 items to record the extent of current dysfunctional behaviors. Ratings are typically based on severity, using a scale from "none" to "very strong," with each item scored from 0 to 4, where 0 indicates no problem and 4 indicates the most severe level. The total score is the sum of all item scores, with higher scores reflecting greater severity of symptoms.
Empathy differentiation index | At baseline, week 4, and week 8
  The Interpersonal Reactivity Index-C (IRI) is a tool used to measure individual differences in empathy. The scale consists of 28 items that encompass four relatively independent dimensions: fantasy, empathic concern, perspective taking, and personal distress. Ratings are typically based on a scale from 0 to 4, corresponding to "does not apply at all," "partially applies," "somewhat applies," "mostly applies," and "fully applies." The scores for each dimension are calculated by summing the ratings of the relevant items and averaging them, with higher scores indicating a stronger empathetic ability in that dimension.
Callous-Unemotional traits assessment index | At baseline, week 4, and week 8
  The Inventory of Callous-Unemotional (ICU) is used to measure callous-unemotional traits. The scale consists of 24 items that assess three dimensions: Callousness, Uncaring, and Unemotional. Each statement is rated on a scale from "does not apply at all" to "applies completely," with scores ranging from 0 to 3 for each item. A higher total score indicates a more pronounced presence of traits in that dimension.
Athens insomnia evaluation index | At baseline, week 4, and week 8
  The Athens Insomnia Scale (AIS) is used to evaluate insomnia. It consists of 8 items, with each item rated on a scale from "no problem" to "mild," "moderate," and "severe or almost no sleep," corresponding to scores of 0 to 3. Respondents rate their sleep quality based on the severity of their insomnia symptoms. The total score of the AIS is the sum of the scores of all entries. A higher total score indicates poorer sleep quality.
Autism spectrum traits assessment index | At baseline, week 4, and week 8
  The Autism Spectrum Quotient-10 (AQ-10) is a simplified self-report screening tool designed to assess the presence of traits associated with Autism Spectrum Disorder (ASD). The scale consists of 10 items, each rated on a 4-point scale ranging from "strongly agree" to "strongly disagree," with scores assigned as 1, 1, 0, and 0. A higher total score indicates a greater likelihood of the individual exhibiting characteristics of Autism Spectrum Disorder.
Empathic ability assessment index | At baseline, week 4, and week 8
  The Empathy Quotient-10 (EQ-10) is a brief self-assessment tool designed to evaluate an individual's empathic ability. The scale consists of 10 items that assess the individual's skills in recognizing, understanding, and responding to the emotions of others. Each item is rated on a scale of 0 to 2 based on the responses "strongly agree," "slightly agree," "slightly disagree," and "strongly disagree," with scores assigned as 2, 1, 0, and 0. A lower total score indicates a poorer level of empathic ability.
Systemizing cognitive style index | At baseline, week 4, and week 8
  The Systemizing Quotient-10 (SQ-R-10) is a self-report measure designed to assess an individual's systemizing cognitive style. This simplified version is based on the more comprehensive Systemizing Quotient-Revised (SQ-R) questionnaire and consists of 10 items aimed at quickly evaluating an individual's propensity for systemizing. Each item is rated on a scale of 0 to 2 based on the responses "strongly agree," "slightly agree," "slightly disagree," and "strongly disagree," with scores assigned as 2, 1, 0, and 0. A higher total score indicates a greater presence of traits associated with autism.
Sensory sensitivity assessment scale | At baseline, week 4, and week 8
  The Sensory Perception Quotient (SPQ) is a self-report tool designed to quantify basic sensory sensitivity in adults. The scale consists of 10 items, each rated on a 4-point scale ranging from "strongly agree" to "strongly disagree," with scores assigned as 3, 2, 1, and 0. A higher total score indicates greater sensory sensitivity.
Behavioral inhibition and activation systems index | At baseline, week 4, and week 8
  The Behavioral Inhibition and Activation Systems Scale (BIS/BAS Scale) is used to measure an individual's behavioral inhibition and activation systems based on reinforcement sensitivity theory. This scale consists of 24 items, divided into two systems: the Behavioral Inhibition System and the Behavioral Activation System, which further includes dimensions such as reward responsiveness, drive, and pleasure-seeking. Scoring employs a 4-point scale ranging from "strongly agree" to "strongly disagree," corresponding to scores of 1 to 4. The total score is the sum of all item scores, with higher scores typically reflecting greater activity in the behavioral activation system, while lower scores indicate a tendency toward behavioral inhibition.
Adult Self-Report (ASR) psychopathology index | At baseline, week 4, and week 8
  The Adult Self-Report (ASR) is part of the Achenbach System, designed to assess adaptive functioning and psychopathology (Achenbach and Rescorla, 2003; Achenbach et al., 2017). The ASR includes eight syndrome scales, with internalizing problems comprising Anxious/Depressed (18 items), Withdrawn (9 items), and Somatic Complaints (12 items), while externalizing problems consist of Aggressive Behavior (15 items), Rule-breaking Behavior (14 items), and Intrusive Behavior (6 items). Other syndrome scales include Attention Problems (15 items) and Thought Problems (10 items), along with 21 additional items that do not fit any syndrome. The total score on the ASR is based on all problem items (120 items in total) and reflects the total problems score for adult psychopathology. Scoring is categorized into three levels: "not true" (0 points), "somewhat or sometimes true" (1 point), and "very true or often true" (2 points).

OTHER OUTCOMES:
Plasma metabolite levels assessment | At baseline, week 4, and week 8
  The levels of metabolites in plasma will be detected and quantified using a comprehensive Metabolomics detection approach. This method involves analyzing small-molecule chemical compounds found in plasma, providing a broad snapshot of the metabolic state of an organism at the given time points.
Safety evaluation SAFTEE indicator | At baseline, week 4, and week 8
  This scale is the most common safety assessment tool used in clinical trials to assess whether participants experienced side effects or unexpected adverse events during the course of the study. The SAFTEE-GI (General inquiry) version was used in this study, which included detailed inquiry on whether subjects had physical or psychological problems in a specific period of time, occurrence time, duration, occurrence frequency, current status, etc., so as to identify adverse reactions of subjects in the course of clinical trials in a timely manner.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Ou, Doctor, Study Chair — Central South University
Locations (1):
- Department of Psychiatry, Xiangya Second Hospital, Central South University, Changsha, Hunan, China